CLINICAL TRIAL: NCT05637658
Title: The Effect of Aerobic Exercise on Nomophobia and Anxiety in Nomophobic University Students
Brief Title: The Effect of Aerobic Exercise on Nomophobia and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karataynomofobia
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No application will be made to the participants in the control group.
- Exercise group (Experimental): Participants will perform aerobic exercise 3 times a week at an intensity of 60-80% of age-adjusted maximal heart reserve on the treadmill and bicycle ergometer for 4 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — aerobic exercise
  Arms: Exercise group

SUMMARY:
It was aimed to examine the effect of aerobic exercise on nomophobia and anxiety in nomophobic university students.

DETAILED DESCRIPTION:
It was aimed to examine the effect of aerobic exercise on nomophobia and anxiety in nomophobic university students. There is no study in the literature examining the relationship between aerobic exercise and nomophobia in young people. Since our study will be the first to investigate the subject, we foresee that it is scientifically important and will shed light on future studies. In addition, national or international publications are planned after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who scored above 22 points on the Beck anxiety scale and 60 points or higher on the nomophobia scale

Exclusion Criteria:

* any condition that may prevent the participant from exercising

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nomophobia score at four weeks | baseline and 4 weeks
  The Nomophobia scale, a 7-point Likert scale consisting of 20 questions developed by Yildirim & Correia, was used to evaluate the nomophobia levels of the participants.Those with a total scores less than 20 did not have nomophobia, 21-59 had mild,60-99 had modarate,and 100-140 had extreme nomophobia

SECONDARY OUTCOMES:
Change from baseline in anxiety score at four weeks | baseline and 4 weeks
  The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in adolescents and adults ages 17 and older.A maximum of 63 points can be obtained from the scale.Less than 21 points indicates mild anxiety, 22-35 points moderate and above 36 points severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided